CLINICAL TRIAL: NCT01923987
Title: Multicenter Phase II Study of Short Course Radiotherapy Followed by Intensive Chemotherapy With Delayed Surgery for Rectal Cancer With Synchronous Distant Metastasis
Brief Title: Short Course Radiotherapy Followed Intensive Chemotherapy With Delayed Surgery for Rectal Cancer With Synchronous Distant Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); Gachon University Gil Medical Center (Other); Catholic University of Korea, Yeouido St. Mary's Hospital (Unknown); Pusan National University Yangsan Hospital (Other); Gangnam Severance Hospital (Other); Severance Hospital (Other); Wonju Severance Christian Hospital (Other); Chungnam National University Hospital (Other); Dongtan Sacred Heart Hospital (Other); The Koreran Society of Coloproctology (Unknown); The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Mi Moon, Korea Cancer Center Hospital, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-1208-001-002; KCT0000525 (Registry Identifier: Clinical Research Information Service); K-1208-001-002 (Other: Korea Institute of Radiological and Medical Sciences IRB)
Record Dates: First submitted 2013-08-07; First posted 2013-08-16 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Rectal Cancer; Liver Metastasis; Lung Metastasis
Keywords: Short course radiotherapy; Modified FOLFOX6; Delayed surgery; Rectal cancer; Synchronous metastasis; Liver metastasis; Lung metastasis
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Folfox protocol; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCRT/ChemoTx with Delayed Surgery (Experimental): Short course radiotherapy (25 Gy in 5 fractions) followed by intensive chemotherapy, compromising of FOLFOX of FOLFIRI (+-Bevacizumab or Cetuximab), with delayed surgery for rectal cancer with synchronous distant metastasis
  Interventions: Radiation: Short Course Radiotherapy; Drug: Chemotherapy; Procedure: Delayed Surgery

INTERVENTIONS:
Radiation: Short Course Radiotherapy — Radiotherapy to tumor and draining lymph node with 25 Gy in 5 fractions within 5 working days
  Other Names: Upfront Short-Course Radiotherapy
Drug: Chemotherapy — * Oxaliplatin 85 mg/m2 IV over 2 hrs on Day 1
  * Irinotecan 180 mg/m2 IV over 30-90 mins on Day 1
  * Leucovorin 400 mg/m2 IV over 2 hrs on Day 1 and 2
  * 5-fluorouracil bolus 400 mg/m2 IV push on Day 1 and 2 (or 5-fluorouracil infusion 600 mg/m2 IV continuous infusion over 22 hrs).
  * Bevacizumab 5 mg/kg IV over 90 mins on Day 1
  * Cetuximab (only for patients with K-ras wild type and positive EGFR mutation) 400 mg/m2 IV over 2 hrs on Day 1, and 250 mg/m2 IV over 1 hr on Day 8, 15, 22, 29, and 36.
  * FOLFOX or FOLFIRI (+-Bevacizumab ) repeats every 14 days for up to 3 courses. Cetuximab repeats every week for up to 6 courses
  * Postoperative FOLFOX or FOLFIRI (+-Bevacizumab or Cetuximab) for up to 9 cycles (total 12 cycles)
  Other Names: FOLFOX or FOLFIRI (+-Bevacizumab or Cetuximab)
Procedure: Delayed Surgery — If primary tumor and metastases is resectable after FOLFOX or FOLFIRI (+-Bevacizumab or Cetuximab) of 3 cycles, patients have surgical resection (and/or radiofrequency ablation to metastases).
  Other Names: Total (or Tumor-specific) mesorectal excision

SUMMARY:
Radical treatment of primary rectal cancer with synchronous distant metastases includes surgical resection of primary and metastatic lesion. However, primary rectal cancer in case of metastasized disease are often locally advanced disease and need downsizing before surgery. It is reported that pelvic recurrence rates and distant metastasis rates outside liver are 30~35% and 60%, respectively. Therefore, combined treatment with radiotherapy and chemotherapy is used. However, the sequence of treatment modalities is not yet definitely established and preoperative chemoradiotherapy and surgical resection is accepted as an option of treatment. Conventional long course chemoradiotherapy delays administration of full-dose chemotherapy, and metastatic lesion can be progressed during chemoradiotherapy. In present study, we evaluate the efficacy of short course radiotherapy (SCRT) followed by full-dose chemotherapy with delayed surgical resection of the primary tumor and metastases.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of rectum
* Lower margin of tumor within 12 cm from anal verge
* Clinically locally advanced (T3-4 or N1-2) disease
* Potentially resectable and synchronous distant metastases in liver and/or lung. The resectability of metastatic lesions is determined by size, number, location, general condition, liver function, and lung function.
* Over 18 years
* Eastern Cooperative Oncology Group performance status 0-2
* Proper organ function (Hemoglobin ≥ 10 g/dl, Absolute neutrophil count (ANC) ≥ 1,500/mm3, Platelet ≥ 100,000/mm3, Creatinine ≤ 1.5 mg/dl, Clearance of creatinine >50 ml/min using Cockcroft-Gault formula, Bilirubin ≤ 1.5 x upper limit of normal (ULN), Liver enzyme (Aspartate aminotransferase/Alanine transaminase/Alkaline phosphatase) ≤ 2.5 x ULN)
* Subject who should sign on the informed consent form before participate the trial.

Exclusion Criteria:

* Metastases in other organ except liver or lung
* History of other type of malignancies within 3 years other than non-melanoma of the skin or carcinoma in situ of cervix
* Hereditary colorectal cancer (FAP, HNPCC, and etc)
* Bowel obstruction or impending bowel obstruction
* Uncontrolled severe illness, unsuitable to chemoradiotherapy (within 6 months, myocardial infarct, unstable angina, heart failure, uncontrolled arrhythmia, uncontrolled epilepsy, central nervous system disease, psychological disorder, and etc)
* Subject pregnant or breast feeding, or incapable of appropriate contraception
* Unresected synchronous colorectal cancer
* History of prior pelvic radiotherapy
* History of prior chemotherapy for colorectal cancer
* Great surgery within 4 week before study enrollment
* Participant in other trial within 4 week before study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2012-08; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | Expected average of 12 weeks (after resection)
  R0 resection rate of primary and metastatic lesions

SECONDARY OUTCOMES:
Overall survival rate | 2 years
  From the first date of radiotherapy to the date of death or last follow-up
Progression free survival rate | 2 years
  From the first date of radiotherapy to the date of first failure or last follow-up
Tumor regression grade | Just after resection & pathologic report
  Tumor regression grade of primary lesion
Toxicity | 1 year
  Adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Sun Mi Moon, MD, PhD, Principal Investigator — Korea Cancer Center Hospital
Locations (2):
- South Korea (2):
  - Kyung Hee University Gangdong Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No